CLINICAL TRIAL: NCT06620926
Title: Impact of IDH Mutation and Adjuvant Chemo(radio)therapy on Survival Outcome in Grade II/III Astrocytoma
Status: Completed | Type: Observational
Sponsor: asmaa salama ibrahim (Other)
Responsible Party: Sponsor-Investigator, asmaa salama ibrahim, Resident physician of gastroenterology, Suez Canal University
Organization: Suez Canal University (Other)
Other Study IDs: A1997
Record Dates: First submitted 2024-09-28; First posted 2024-10-01 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Astrocytoma; Astrocytic Tumors; Astrocytoma of Brain
Keywords: chemotherapy; survival; Astrocytoma; Wild IDH
MeSH Terms: conditions — Astrocytoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients having astrocytoma with IDH mutant-type
  Interventions: Other: IDH mutant-type
- Patients having astrocytoma with IDH wild-type
  Interventions: Other: IDH wild-type

INTERVENTIONS:
Other: IDH mutant-type — The first arm had IDH mutant-type, then stratified according to the treatment modality they received: adjuvant chemotherapy, adjuvant radiotherapy, adjuvant chemoradiotherapy.
  Groups: Patients having astrocytoma with IDH mutant-type
Other: IDH wild-type — The second arm had IDH mutant-type, then stratified according to the treatment modality they received: adjuvant chemotherapy, adjuvant radiotherapy, adjuvant chemoradiotherapy.
  Groups: Patients having astrocytoma with IDH wild-type

SUMMARY:
This study looked at a type of brain tumor called astrocytoma and how specific genetic changes like IDH mutations affect patients outcomes. Recent studies found that people with IDH-mutated astrocytomas tend to live longer and have better survival rates compared to those without these mutations. One reason for this is that IDH-mutated tumors usually grow more slowly and are less aggressive. These findings suggest that testing for IDH mutations could help doctors make more personalized treatment plans for patients, which may lead to better results. However, larger studies are needed to confirm these observations. the investigators used the Surveillance, Epidemiology and End Results (SEER) database to obtain the data of 811 patients with grade II/III astrocytoma. The data are publicly available and no consent or ethical approval is needed for this study. The clinicopathological data of patients, including the age, gender, race, IDH status (mutant/wild), astrocytoma type (diffuse/anaplastic), surgery (tumor destruction, Local excision, partial, radical, total gross resection, Surgery), radiation (Beam radiation, Radioactive implants including brachytherapy, Radioisotopes, Combination of beam with implants or isotopes, Radiation, method or source not specified), chemotherapy, vital status, and survival months, were extracted. Patients were sub-grouped according to the IDH type into IDH mutant-type and wild-type. with further stratification according to the treatment modality into three groups: adjuvant chemotherapy, adjuvant radiotherapy, and combined adjuvant chemoradiotherapy. The Observed survival and cause-specific survival were calculated using SEER*stat software version 8.4.3 and SPSS version 25 was used for survival analysis. Significance was achieved at 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients were selected only if they had astrocytoma with malignant behavior
* Grade II-III astrocytoma
* First primary tumor with sequence 0 or 1
* Had surgical intervention (tumor destruction, Local excision, partial, radical, total gross resection, Surgery)

Exclusion Criteria:

* unknown survival time
* patients with unknown age
* death certificate only and autopsy only cases

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with grade II/III astrocytoma with malignant behavior. The investigators sub-grouped the data according to the IDH mutation type into two groups: IDH wild-type and IDH-mutant type with further stratification according to the treatment modalities the patients received: adjuvant chemotherapy, adjuvant radiotherapy and adjuvant chemoradiotherapy; following any surgical intervention (tumor destruction, Local excision, partial, radical, total gross resection, Surgery)
Sampling Method: Probability Sample
Enrollment: 811 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
The 2-year relative survival and 2-year observed survival of grade II/III astrocytoma with IDH mutation | from Jan, 2018 till Dec, 2020

SECONDARY OUTCOMES:
The 2-year relative survival of different treatment with modalities chemo(radio)therapy among both groups: IDH wild type and IDH mutant type astrocytoma | Jan, 2018 till Dec, 2020

CONTACTS AND LOCATIONS:
Overall Officials: Asmaa Ellaithy, MD, Principal Investigator — Suez Canal University
Locations (1):
- Suez Canal University, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
The data is publicly available through SEER database

REFERENCES:
- [Derived] Hamad M, Ali MA, Hamouda E, Hamouda H, Ali N, Al-Shaikh B, Ellaithy A. Impact of IDH mutation and adjuvant chemo(radio)therapy on survival outcome in grade II/III astrocytoma: a retrospective cohort study based on SEER database. Ann Med Surg (Lond). 2025 Mar 20;87(4):1846-1851. doi: 10.1097/MS9.0000000000003172. eCollection 2025 Apr. PMID 40212132